CLINICAL TRIAL: NCT06408259
Title: A Phase 3, Multicenter, Double-blind, Active-controlled Study to Evaluate the Efficacy, Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Oral Ozanimod Compared to Oral Fingolimod in Children and Adolescents With Relapsing Remitting Multiple Sclerosis
Brief Title: Study to Evaluate the Effectiveness and Safety of Ozanimod Compared to Fingolimod in Children and Adolescents With Relapsing Remitting Multiple Sclerosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM047-050; 2022-501332-42 (Registry Identifier: EU Trial Number); U1111-1281-5433 (Registry Identifier: UTN)
Record Dates: First submitted 2024-04-25; First posted 2024-05-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis; Relapsing-Remitting; Ozanimod; Zeposia®
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — ozanimod; Fingolimod Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ozanimod (Experimental)
  Interventions: Drug: Ozanimod; Other: Placebo
- Fingolimod (Active Comparator)
  Interventions: Drug: Fingolimod; Other: Placebo

INTERVENTIONS:
Drug: Ozanimod — Specified dose on specified days
  Arms: Ozanimod
Drug: Fingolimod — Specified dose on specified days
  Arms: Fingolimod
Other: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the effectiveness, safety, tolerability, drug levels and drug effects of ozanimod compared to fingolimod in children and adolescents with relapsing remitting multiple sclerosis (RRMS).

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of multiple sclerosis (MS) as defined by the 2017 revision of the McDonald Criteria with a relapsing remitting course of disease.
* Meets at least 1 of the following criteria for disease activity:

  i) At least 1 MS relapse/attack in the previous year prior to screening.

ii) At least 2 MS relapses/attacks in the previous 2 years prior to screening.

iii) Evidence of 1 or more gadolinium-enhancing (GdE) lesions on magnetic resonance imaging (MRI) within 6 months prior to baseline (including screening MRI).

- Has an Expanded Disability Status Scale (EDSS) score of 0 to 5.5, both inclusive.

Exclusion Criteria:

* Diagnosis of progressive forms of MS.
* Active or chronic disease of the immune system other than MS.
* Clinically relevant cardiovascular, hepatic, neurological other major systematic disease.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 194 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2031-04-11 (Estimated); Study Completion 2036-07-13 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate (ARR) | Up to 2 years

SECONDARY OUTCOMES:
Proportion of participants who did not have a confirmed relapse | At 12 and 24 months
Number of gadolinium enhancing (GdE) T1 lesions | At month 6 and month 12
Number of new or newly enlarging hyperintense lesions on T2 magnetic resonance imaging (MRI) sequences | At 6, 12, 18, and 24 months
Incidence of treatment-emergent adverse events (TEAEs) over the treatment period and over the post-treatment follow-up period | Up to 87 months
Incidence of adverse event of special interests (AESIs) over the treatment period and over the post-treatment follow-up period | Up to 87 months
Adverse events (AEs) leading to discontinuation over the treatment period and over the post-treatment follow-up period | Up to 87 months
Steady state plasma concentrations of ozanimod | At day 90
Steady state plasma concentrations of the primary active metabolite CC112273 | At day 90
Change from baseline pharmacodynamics (PD) biomarkers of absolute lymphocyte count | At day 90 and throughout the study up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (33):
- United States (12):
  - Local Institution - 0114, Loma Linda, California
  - University of California Davis Health, Sacramento, California
  - University of South Florida, Tampa, Florida
  - Local Institution - 0093, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Local Institution - 0047, Louisville, Kentucky
  - Local Institution - 0131, New Brunswick, New Jersey
  - Local Institution - 0132, Teaneck, New Jersey
  - Local Institution - 0091, Cincinnati, Ohio
  - Local Institution - 0092, Portland, Oregon
  - Local Institution - 0133, El Paso, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Royal Children's Hospital, Melbourne, Victoria, Australia
- Italy (4):
  - University of Naples Federico II, Napoli, Campania
  - Ospedale San Raffaele, Milan, Lombardy
  - Local Institution - 0081, Milan, Lombardy
  - Neurological Center Of Latium, Rome, Roma
- Local Institution - 0078, Mexico City, DIF, Mexico
- Uniwersytecki Szpital Kliniczny w Poznaniu, Poznan, Greater Poland Voivodeship, Poland
- Portugal (4):
  - 2Ca Braga, Braga
  - Unidade Local de Saúde de Coimbra, E.P.E., Coimbra
  - Centro Hospitalar de Lisboa Central, Lisbon
  - Local Institution - 0102, Porto
- Local Institution - 0134, Caguas, Puerto Rico
- Romania (2):
  - Spitalul Clinic de Copii Doctor Victor Gomoiu, Bucharest, București
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest, București
- Spain (5):
  - Local Institution - 0096, Esplugues de Llobregat, Barcelona [Barcelona]
  - CHUVI- Hospital Alvaro Cunqueiro, Vigo, Pontevedra [Pontevedra]
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- National Taiwan University Hospital, Taipei, Taiwan
- Ondokuz Mayıs Universitesi, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html